CLINICAL TRIAL: NCT05071014
Title: A Phase 1 Study of Pembrolizumab Plus Cryoablation in Patients With Unresectable Mesotheliomas
Brief Title: A Study of Pembrolizumab and Cryoablation in People With Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-342
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer; Unresectable Mesothelioma
Keywords: Pembrolizumab; Cryoablation; 21-342
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This clinical trial will be designed as a single-arm, single-institution study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab followed by cryoablation (Experimental): The treatment will consist of 1 cycle of pembrolizumab (200mg/flat dose) intravenously followed by cryoablation of an ablation index lesion 1-7 days prior to the start of cycle 2. Pembrolizumab will be continued for up to 24 months, until disease progression, or intolerable toxicity. Treatment beyond progression at discretion of the treating physician and Study PI. There will be a research biopsy within 1 week of cycle 5 start and an optional biopsy at end of treatment and/or progression of disease.
  Interventions: Drug: Pembrolizumab; Procedure: Image-guided cryoablation

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab: 200mg/dose delivered by IV infusion
Procedure: Image-guided cryoablation — Cryoablation will be used to treat a designated lesion with preference given to a lesion that is symptomatic or at risk of causing symptoms. Per institutional standards, complete ablation of the lesion will be attempted.

SUMMARY:
The researchers are doing this study to find out whether the combination of pembrolizumab and cryoablation is a safe treatment that causes few or mild side effects in people with mesothelioma. The researchers will also look at whether the combination of pembrolizumab and cryoablation is effective against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to provide written informed consent for the trial
* Patient age ≥ 18 at time of consent
* Unresectable mesothelioma
* Histologically or cytologically confirmed unresectable mesothelioma (pleural or peritoneal) as assessed by dedicated collaborators from the Departments of Pathology and Surgery.
* At least one prior line of systemic therapy. Prior immunotherapy (as defined as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4)) is allowed if it did not contain pembrolizumab and was not the most recent therapy, unless last treated ≥ 1 year from trial enrollment
* Multifocal disease with at least one mRECIST v1.1 evaluable lesion medically safe/feasible for palliative cryoablation, as determined by the treating Interventional Radiologist, and at least one other mRECIST v1.1 measurable lesion to be monitored that will not undergo cryoablation
* Agree to undergo research biopsy of the ablated lesion ± non-ablated lesion at the time of cryoablation and prior to cycle 5 if deemed medically safe and feasible
* Informed consent to 12-245 and 06-107
* Karnofsky Performance Score (KPS) ≥ 70%
* Adequate organ function defined as:

  * Absolute Neutrophil Count ≥ 1.5K/mcL
  * Platelet count ≥ 100K/mcL
  * Adequate renal function as defined as Creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 45ml/min (as calculated by Cockcroft-Gault Formula)
  * Hemoglobin ≥ 9g/dL (prior transfusion permitted if not within 7 days or enrollment )
  * Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range
  * AST and ALT levels ≤ 3.0 × ULN or AST
* If the patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* If of childbearing potential, must be willing to use highly effective mode of contraception for at least one month prior, during, and for 2 months after the end of active therapy

Exclusion Criteria:

* Currently participating and receiving another study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Continuous supplemental oxygen use
* Active autoimmune disease that might deteriorate when receiving an immuno- stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* Known prior severe hypersensitivity to pembrolizumab or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3)
* Patient who rapidly progressed on prior immunotherapy, as determined by the treating physician or Primary Investigator, are not eligible
* Prior cytotoxic/immunologic systemic therapy within 4 weeks prior to study Day 1 or has not recovered (i.e., ≥ Grade 1 at baseline) from adverse events due to a previously administered agent (excluding Grade 2 neuropathy)
* Comorbidities or prior conditions:

  * Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
  * Prior organ transplantation including allogenic stem-cell transplantation
  * Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early stage prostate cancer, or in situ cervical cancer after definitive treatment
  * Known history of HIV or known acquired immunodeficiency syndrome.
  * Active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection at screening
  * Evidence of interstitial lung disease or active, non-infectious pneumonitis.
  * Clinically significant (i.e., active) cardiovascular disease as determined by anesthesiology and/or Interventional Radiology which would preclude the safe execution of cryoablation
* Concomitant use of the following medications

  * Any investigational anticancer therapy.
  * Any concurrent chemotherapy, immunotherapy, or biologic therapy. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
  * Systemic anticoagulation which cannot safely be held for cryoablation/biopsies; length of anticoagulation pause will be determined by Interventional Radiology as per standard of care practices.
  * Immunosuppressive medications including, but not limited to systemic corticosteroids (>10 mg/day prednisone or equivalent), methotrexate, azathioprine, and tumor necrosis factor alpha (TNF-α) blockers. Use of steroids for contrast allergies is acceptable. In addition, use of inhaled and intranasal corticosteroids is permitted.
* Pregnant women or women who are breastfeeding or of childbearing potential and not using a highly effective method of birth control for at least one month prior to enrollment. If the risk of contraception exists, male and female subjects must use highly effective contraception throughout the study and for at least 60 days after last pembrolizumab treatment.

  * Highly effective contraception includes either 2 barrier methods (diaphragm, condom by the partner, copper intrauterine device, sponge, or spermicide), or 1 barrier method and 1 hormonal method (any oral, subcutaneous, intrauterine, or intramuscular registered and marketed contraceptive agent that contains an estrogen and/or a progesterone agent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
number of patients with an adverse event (AE) defined as any grade 3 or higher non-hematologic toxicity | within 12 weeks of cryoablation
  Adverse event severity is graded per NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Offin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm